CLINICAL TRIAL: NCT00039182
Title: A Phase II Study of Oral EGFR Tyrosine Kinase Inhibitor OSI-774 (NSC-718781) in Patients With Malignant Pleural Mesothelioma
Brief Title: Erlotinib in Treating Patients With Malignant Mesothelioma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02466; SWOG-S0218; U10CA032102 (NIH); CDR0000069360 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. This phase II trial is studying how well erlotinib works in treating patients with malignant mesothelioma of the lung

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 1-year survival rate in patients with unresectable malignant pleural mesothelioma treated with erlotinib.

II. Determine the response rate in patients with measurable disease treated with this drug.

III. Determine the frequency and severity of toxic effects of this drug in these patients.

IV. Measure epidermal growth factor receptor (EGFR) expression, EGFR gene amplification, and other activation products in the EGFR signaling pathway in tumor samples and correlate with clinical outcomes in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 2 years and then annually for 1 year.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 14-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant pleural mesothelioma

  * Epithelial
  * Sarcomatous
  * Biphasic
* Measurable or nonmeasurable disease
* Not amenable to extrapleural pneumonectomy
* No known CNS metastases
* Performance status - Zubrod 0-1
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 1.5 times ULN (5 times ULN if liver involvement of tumor)
* Creatinine no greater than 2 times ULN
* No gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No active peptic ulcer disease
* No intractable nausea or vomiting
* Must be able to swallow and/or receive enteral medications via gastrostomy feeding tube
* No known history of the following:

  * Dry eye syndrome
  * Sjogren's syndrome
  * Keratoconjunctivitis sicca
  * Exposure keratopathy
  * Fuch's dystrophy
  * Other active disorders of the cornea
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No HIV-positive patients receiving combination antiretroviral therapy
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer that is in complete remission
* No prior biologic therapy for this tumor
* No prior chemotherapy for this tumor
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* See Disease Characteristics
* At least 4 weeks since prior major surgery (e.g., thoracotomy or laparotomy), excluding minor surgeries (e.g., mediastinoscopy, thoracoscopy, or minor biopsies)
* Recovered from prior surgery
* No prior surgical procedures affecting absorption
* No prior investigational anticancer agents for this tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-05; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 1 year
  Erlotinib hydrochloride will not be of further interest if the true one-year survival rate is 35% or less, but of considerable interest if 55% or more.
RECIST response rate | Up to 3 years
Association between EGFR expression with survival and response | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garland, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States